CLINICAL TRIAL: NCT01901705
Title: A Study of Topical Indigo Naturalis Treatment in Patients With Mild to Moderate Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMR101-IRB1-261; DMR101-IRB1-261 (Other: China Medical University Hospital)
Record Dates: First submitted 2013-05-09; First posted 2013-07-17 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Psoriasis
Keywords: Psoriasis; Indigo Naturalis; chinese medicine
MeSH Terms: conditions — Psoriasis | interventions — Qingdai compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indigo (Active Comparator): The Indigo naturalis ointment will be provided and patients are instructed to use it twice daily for 8 weeks or achieve completely skin clearing whichever comes first.
  Interventions: Drug: Indigo naturalis ointment
- Placebo (Placebo Comparator): The Placebo will be provided and patients are instructed to use it twice daily for 8 weeks or achieve completely skin clearing whichever comes first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indigo naturalis ointment — The Indigo naturalis ointment was composed of a 1:10 mixture of Indigo naturalis powder and a vehicle consisting of Vaseline: microcrystalline wax: olive oil (5:6:9 ratio)
  Arms: Indigo
Drug: Placebo — The placebo was a mixture of blue dye powder (54.8% Indigo carmine aluminum lake [Blue #32] and 45.2% Allura Red AC aluminum lake [Red #40] powders), Vaseline, microcrystalline wax, and olive oil.
  Arms: Placebo

SUMMARY:
Psoriasis is a common, chronic skin disease for which only remissive, as opposed to curative, treatments are available. Traditional Chinese medicine is one of the most frequently chosen alternative therapies in China and Taiwan, and psoriasis has been treated for centuries with topical and oral herbal preparations. Topical indigo naturalis ointment has been reported to exhibit potential anti-psoriatic efficacy. The study objective is to investigate pharmacological effect and explore targeting mechanisms of Traditional Chinese Medicine (TCM) Indigo Naturalis topical ointment as a single treatment agent in Chinese subjects with mild to moderate plaque-type Psoriasis.

This was a single site, randomized, double-blinded, placebo controlled study of topical indigo naturalis vs. vehicle alone (placebo) to treat mild to moderate plaque-type psoriasis during an 8-week period. Pharmacological effect will be evaluated by biomarker evaluation and clinical evaluation. The trial was conducted at the China Medical University Hospital (CMUH), Taichung, Taiwan. All patients provided written informed consent before inclusion in the study. The study protocol was approved by the institutional review board (IRB) of CMUH.

DETAILED DESCRIPTION:
Estimated enrollment:

Total of 24 subjects:

mild to moderate psoriasis patients will be randomized into treatment group (n=16) placebo group (n=8)

Study evaluation:

A baseline and end of the study evaluation on the patients will be performed, including physical examination, hemogram and blood biochemical analysis (including glutamic-oxaloacetic transaminase, glutamic-pyruvic transaminase, and creatinine measurement). The baseline and end of the study of total body surface area involvement and Psoriasis Area Severity Index (PASI), PGA, OTPSS scores will be also calculated.

ELIGIBILITY:
Inclusion Criteria:

* men or women at ages between 20 - 65 years old with at least 6 months diagnosis of moderate to mild plaque-type psoriasis who have a screening and at time of study agent treatment Psoriasis Global Assessment (PGA)=2-3, and have under 20% of their total body surface area (BSA) involved. , with a target plaque for at least 4 sq cm
* In good general health, as evidenced by physical examination, and hematology and blood chemistry tests within normal ranges with the exception of liver function test value <=1.5ULN
* If of childbearing age, agreement to continue using birth control measures for the duration of the study
* Patients who agreed to participate and signed the consent form
* Patients who agreed to return for follow-up visits and provide all required biopsies.

Exclusion Criteria:

* Currently have non-plaque forms of psoriasis (e.g., erythrodermic, guttate, or pustular psoriasis), or rebound or flare of chronic plaque psoriasis
* Currently or had history of psoriatic arthritis
* Have current drug-induced psoriasis (e.g., a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium).
* Are pregnant, nursing, or planning pregnancy (both men and women) while enrolled in the study.
* Have used any biologic within the previous 3 months or 5 times the half-life of the biologic, whichever is longer
* Have received phototherapy or any systemic treatment that could affect psoriasis (including, but not limited to, (eg, retinoids, methotrexate, cyclosporine, psoralens, sulfasalazine, hydroxyurea, fumaric acid derivatives, herbal treatment or traditional Chinese medicine) within 4 weeks of receiving study treatment
* Have used topical treatment that could affect psoriasis (eg. corticosteroid tazarotene, and tacrolimus, tar, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, topical traditional Chinese medicines) within 2 weeks of receiving study treatment
* Have used any systemic immunosuppressants (eg, MTX, azathioprine, cyclosporine, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, and tacrolimus) within 4 weeks of receiving study treatment
* Are currently receiving lithium, antimalarials, or intramuscular gold, or have received lithium, antimalarials, or intramuscular gold within 4 weeks of receiving study treatment
* Positive screening tests for HIV, hepatitis B surface antigen, or hepatitis C antibody
* A history of alcohol or other drug abuse
* Clinically significant laboratory abnormality in blood, renal function, or liver function
* A history of sensitivity to Chinese herbs, olive oil, yellow wax, or petroleum jelly
* Have current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Be participating in another trial using an investigational agent or procedure.
* Any other conditions that in the view of investigator, the subject should not be enrolled.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Overall Target Plaque Severity Score at 8 weeks | Baseline and at 8 weeks
  OTPSS(Overall Target Plaque Severity Score ) Score Description 0 No evidence of disease (except possible residual discoloration)
  1. *
  2. Mild overall plaque elevation, scaling and/or erythema of the target plaque
  3. *
  4. Moderate overall plaque elevation, scaling and/or erythema of the target plaque
  5. *
  6. Severe overall plaque elevation, scaling and/or erythema of the target plaque
  7. *
  8. Very severe overall plaque elevation, scaling and/or erythema of the target plaque *Grades 1, 3, 5 & 7 are midpoints between the defined grades 0, 2, 4, 6 & 8

CONTACTS AND LOCATIONS:
Overall Officials: Hui man cheng, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital,, Taichung, Taiwan

REFERENCES:
- [Derived] Cheng HM, Wu YC, Wang Q, Song M, Wu J, Chen D, Li K, Wadman E, Kao ST, Li TC, Leon F, Hayden K, Brodmerkel C, Chris Huang C. Clinical efficacy and IL-17 targeting mechanism of Indigo naturalis as a topical agent in moderate psoriasis. BMC Complement Altern Med. 2017 Sep 2;17(1):439. doi: 10.1186/s12906-017-1947-1. PMID 28865459